CLINICAL TRIAL: NCT06812468
Title: Anthropometric Parameters of Pristine Maxillary Anterior Teeth and Facial Index in Correlation With Recurring Esthetic Dental Proportion (RED) by 3D Digital Software
Brief Title: Maxillary Anterior Teeth and Facial Index Parameters in Correlation With Recurring Esthetic Dental Proportion
Acronym: RED
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Souad Mohamed, Demonstrator of oral and dental biology departement, Al-Azhar University
Other Study IDs: RED proportion
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: There is no Disease the Study Focus on Facial Index in Relation to RED
Keywords: RED, Facial index, Teeth measurement
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- 10 female patients: the facial index and the anterior teeth dimensions and the interrelation between them were assessed. Finally the results were correlated with recurring aesthetic dental proportion (RED). Moreover the results were statistically analyzed using the Independent t-test or an equivalent non-parametric test was used for comparison between the two groups, and the Pearson's correlation coefficient (r) test was used for correlating different parameters.
  Interventions: Device: Bellus 3D smart application; Device: Medit i-700 intraoral scanner
- 10 males patients: the facial index and the anterior teeth dimensions and the interrelation between them were assessed. Finally the results were correlated with recurring aesthetic dental proportion (RED). Moreover the results were statistically analyzed using the Independent t-test or an equivalent non-parametric test was used for comparison between the two groups, and the Pearson's correlation coefficient (r) test was used for correlating different parameters.
  Interventions: Device: Bellus 3D smart application; Device: Medit i-700 intraoral scanner

INTERVENTIONS:
Device: Bellus 3D smart application — Bellus3D is a modern multi-digital digicam, 3-D face scanning that captures in an expert grade, complete 3-D face scans with the pressing of an unmarried button in seconds. It takes 10 s to create an excessive decision 3-D face scan. Bellus3D's excessive precision scanning detects the soft tissue parameters and over a hundred facial andmarks. It uses two Infrared structured light VCSEL (vertical-cavity surface-emitting laser) projectors for high-resolution face scanning. The technique of facial scanning by (Bellus3D) and measuring facial index by (Medit) software was performed following manufacture instructions , The patient's head Stabilized and aligned with the center of the face scan software (Bellus 3D) to avoid scan distortion, The head was tilted towards right and then towards left along with the face analog in the scan software combined with upward and downward movement to ensure complete detection and record of facial landmarks. Then the obj 3D file exported to Medit Software.
Device: Medit i-700 intraoral scanner — Medit i-700 intra oral scanner was used to measure the teeth dimensions , it has several advantages including that it can capture up to 70 FPS (FRAMES PER SECOND), which is significantly faster than the previous model. It delivers high image resolution for better quality. The Medit i700 offers a remote control mode and a built-in UV-C disinfection function. In this study a zigzage movement was used which more accurate rout for recording all anterior teeth dimensions and surrounding tissue while scanning. In agreement with a previous study, we started from the posterior left area by scanning the occlusal side, then it proceeded toward the posterior right area by following a zigzag movement when the anterior teeth were scanned. After the occlusal area, the palatal/lingual side was scanned from the right to the left area, and then the buccal side was scanned from the posterior left area to the posterior right one,Then the obj 3D file exported to Medit Software.

SUMMARY:
The goal of this cross-sectional study is to state the inter relation between anthropometric parameters of pristine maxillary anterior teeth and facial index and their correlation with recurring esthetic dental proportion (RED) using 3D digital software (Medit) with intra intraoral scanner.The study comprised of 20 adult out patients with an equal number of males and females who had 20-35 years old.

DETAILED DESCRIPTION:
The research focuses on analyzing the proportions of maxillary anterior teeth in relation to facial measurements, particularly within the Egyptian population. It evaluates how closely these dimensions align with the Recurring Esthetic Dental (RED) proportions, which suggest that the width of anterior teeth should decrease by a constant ratio moving distally. Using advanced digital tools such as the BELLUS 3D face scanner and MEDIT i700 intraoral scanner, the study collected detailed facial and dental measurements from participants to explore the correlation between facial index and tooth dimensions. The sample consisted of 20 participants (10 males and 10 females), with data analyzed using statistical methods to assess symmetry and gender variations in these proportions.). Moreover the results were statistically analyzed using the Independent t-test or an equivalent non-parametric test was used for comparison between the two groups, and the Pearson's correlation coefficient (r) test was used for correlating different parameters.

ELIGIBILITY:
Inclusion Criteria:

1. must be in the same age group (20-35). 2. free of systemically disease (GI, D.M., gastric influx). 3. Free of facial asymmetry. 4. Free of facial trauma or surgeries. 6.Normal Class 1 occlusion. 7. Free from any tooth wear disorder. 8.periodontally healthy without any previous orthodontic treatment. 9. Maxillary anterior teeth free from restoration

-

Exclusion Criteria:

1. History of surgery in the anterior maxillary or mandibular region. 2. Restorations in anterior sextant. 3 pregnant or lactating females. 4. gingival hyperplasia. 5. orthodontic treatment. 6. Facial asymmetry and clefts 7.Smokers patient

-

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyption Population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
parameters of pristine maxillary anterior teeth and facial index in correlation with recurring esthetic dental proportion (RED) | 20 years old to 35years old
  Assessment of facial index and facial forms:the morphological face height (n-gn) was measured as the distance between the nasal root (n: nasion) and the lowest point of the lower border of mandible in the mid-sagittal plane, (gn: gnathion), while the maximum facial width was considered as bizygomatic width (zy-zy)which was measured from the left zygion to the right zygion.All measurements were performed by a 3D face scanning software (BELLUS 3D). the overall facial form was calculated according to the formula FI = FW / FH× 100. Assessment of Maxillary Anterior Teeth Dimensions:The dimensions of Maxillary anterior teeth were measured for each case as: width and length of central, lateral and canines, in both right and left segments and inter canine distance. All dimensions were measured using scans which were taken by MEDIT i700 intraoral scanner.Correlating the results with RED proportion :The formula for determining the ideal width of the central incisor is:CIW =ICW/2 (1+RED+RED2).

CONTACTS AND LOCATIONS:
Overall Officials: Heba A Head of oral and dental biology department, Professor of oral and dental, Study Director — Al-Azhar University; Seham I Lecturer of oral biology, PHD, Study Director — Al-Azhar University
Locations (2):
- Egypt (2):
  - Al Azhar University, Cairo
  - faculty of dentistry, Al azhar University for girls, Nasr City, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in RED proportion. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication, and the data will be made accessible for up to 24 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Gadallah MA, Khamis MM, Abdelhamid AM, Ezzelarab S. Evaluation of the use of different intraoral scanners for auricular prosthetic reconstruction. J Prosthet Dent. 2025 Aug;134(2):513-519. doi: 10.1016/j.prosdent.2023.09.028. Epub 2023 Oct 27. PMID 39492256
- [Background] Dag OD, Dagli I, Kurt A. The influence of different tooth proportions obtained using digital smile design on the perception of smile esthetics. J Esthet Restor Dent. 2024 Mar;36(3):494-502. doi: 10.1111/jerd.13164. Epub 2023 Nov 11. PMID 37950584
- [Background] Fung L, Brisebois P. Implementing Digital Dentistry into Your Esthetic Dental Practice. Dent Clin North Am. 2020 Oct;64(4):645-657. doi: 10.1016/j.cden.2020.07.003. Epub 2020 Aug 12. PMID 32888514
- [Background] Al-Kaisy N, Garib BT. Analysis of the golden proportion and width/height ratios of maxillary anterior teeth in Arab and Kurdish populations. J Prosthet Dent. 2018 Jun;119(6):981-986. doi: 10.1016/j.prosdent.2017.08.017. Epub 2017 Nov 15. PMID 29153745
- [Background] Ahmed N, Halim MS, Aslam A, Ghani ZA, Safdar J, Alam MK. An Analysis of Maxillary Anterior Teeth Crown Width-Height Ratios: A Photographic, Three-Dimensional, and Standardized Plaster Model's Study. Biomed Res Int. 2022 Feb 7;2022:4695193. doi: 10.1155/2022/4695193. eCollection 2022. PMID 35229002
- [Background] Liao P, Fan Y, Nathanson D. Evaluation of maxillary anterior teeth width: A systematic review. J Prosthet Dent. 2019 Sep;122(3):275-281.e7. doi: 10.1016/j.prosdent.2018.10.015. Epub 2019 Apr 5. PMID 30955941
- [Background] Akl MA, Mansour DE, Mays K, Wee AG. Mathematical Tooth Proportions: A Systematic Review. J Prosthodont. 2022 Apr;31(4):289-298. doi: 10.1111/jopr.13420. Epub 2021 Sep 23. PMID 34463403
- [Background] Alaghbari SSA, Mohmmed BSA, Alalwani NNM, Sobhy MM, Qadi KA, Khawaji SA, Mhbob HO, Alsadi FM, Moaleem MMA. Analysis of the Facial Measurements and Dental Arch Dimensions for the Construction of Dental Prostheses among Adult Yemenis. J Contemp Dent Pract. 2023 Aug 1;24(8):595-604. doi: 10.5005/jp-journals-10024-3511. PMID 38193184
- [Background] Wang Y, Song Y, Zhong Q, Xu C. Evaluation of influence factors on the width, length, and width to length ratio of the maxillary central incisor: A systematic review and meta-analysis. J Esthet Restor Dent. 2021 Mar;33(2):351-363. doi: 10.1111/jerd.12606. Epub 2020 Jul 8. PMID 32643266
- [Background] Cinelli F, Piva F, Bertini F, Russo DS, Giachetti L. Maxillary Anterior Teeth Dimensions and Relative Width Proportions: A Narrative Literature Review. Dent J (Basel). 2023 Dec 25;12(1):3. doi: 10.3390/dj12010003. PMID 38248211
- [Background] Radia S, Sherriff M, McDonald F, Naini FB. Relationship between maxillary central incisor proportions and facial proportions. J Prosthet Dent. 2016 Jun;115(6):741-8. doi: 10.1016/j.prosdent.2015.10.019. Epub 2016 Jan 13. PMID 26794701
- [Background] Ward DH. Proportional Smile Design: Using the Recurring Esthetic Dental Proportion to Correlate the Widths and Lengths of the Maxillary Anterior Teeth with the Size of the Face. Dent Clin North Am. 2015 Jul;59(3):623-38. doi: 10.1016/j.cden.2015.03.006. PMID 26140969
- [Background] Jafri Z, Ahmad N, Sawai M, Sultan N, Bhardwaj A. Digital Smile Design-An innovative tool in aesthetic dentistry. J Oral Biol Craniofac Res. 2020 Apr-Jun;10(2):194-198. doi: 10.1016/j.jobcr.2020.04.010. Epub 2020 Apr 18. PMID 32373450
- [Background] Tsuchida Y, Shiozawa M, Handa K, Takahashi H, Nikawa H. Comparison of the accuracy of different handheld-type scanners in three-dimensional facial image recognition. J Prosthodont Res. 2023 Apr 12;67(2):222-230. doi: 10.2186/jpr.JPR_D_22_00001. Epub 2022 Jun 29. PMID 35768278
- [Background] Ellakwa A, McNamara K, Sandhu J, James K, Arora A, Klineberg I, El-Sheikh A, Martin FE. Quantifying the selection of maxillary anterior teeth using intraoral and extraoral anatomical landmarks. J Contemp Dent Pract. 2011 Nov 1;12(6):414-21. doi: 10.5005/jp-journals-10024-1069. PMID 22269230
- [Background] Koidou VP, Chatzopoulos GS, Rosenstiel SF. Quantification of facial and smile esthetics. J Prosthet Dent. 2018 Feb;119(2):270-277. doi: 10.1016/j.prosdent.2017.04.002. Epub 2017 May 26. PMID 28552284
- [Background] Parciak EC, Dahiya AT, AlRumaih HS, Kattadiyil MT, Baba NZ, Goodacre CJ. Comparison of maxillary anterior tooth width and facial dimensions of 3 ethnicities. J Prosthet Dent. 2017 Oct;118(4):504-510. doi: 10.1016/j.prosdent.2016.10.035. Epub 2017 Mar 23. PMID 28343667
- [Background] Yue Z, Luo Z, Hou J, Zhang H. Application of 3D digital smile design based on virtual articulation analysis in esthetic dentistry: A technique. J Prosthet Dent. 2025 Jan;133(1):24-30. doi: 10.1016/j.prosdent.2023.11.014. Epub 2023 Dec 6. PMID 38061939
- [Background] Mangano F, Gandolfi A, Luongo G, Logozzo S. Intraoral scanners in dentistry: a review of the current literature. BMC Oral Health. 2017 Dec 12;17(1):149. doi: 10.1186/s12903-017-0442-x. PMID 29233132
- [Background] Baghiana G, Peter D, Manju V, Babu AS, Krishnan V. Relevance of Recurring Esthetic Dental (RED) proportion and golden proportion among patients attending a tertiary care center at Kochi, Kerala. J Oral Biol Craniofac Res. 2022 Nov-Dec;12(6):890-893. doi: 10.1016/j.jobcr.2022.09.003. Epub 2022 Sep 9. PMID 36277123